CLINICAL TRIAL: NCT04081064
Title: Exploring the Impact of Body Fat Profile, and a Physical Exercise Intervention on Clinical, Metabolic and Molecular Parameters in Qatar Residents With Type 2 Diabetes Mellitus
Brief Title: Impact of Body Composition and Exercise on Clinical, Metabolic and Molecular Parameters in Type 2 Diabetics in Qatar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Hamad Bin Khalifa University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-03-17-0025
Record Dates: First submitted 2019-07-24; First posted 2019-09-06 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes
Keywords: Obese; Non-obese; Qatar
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-obese Qatar residents with type 2 diabetes (Experimental): Newly diagnosed (e.g <5 years) Type 2 diabetics Qatar residents with a body mass index (BMI) of >18.5 and <30.0 kg/m2
  Interventions: Behavioral: 10-week exercise programme based on aerobic interval and resistance training
- Obese Qatar residents with type 2 diabetes (Experimental): Newly diagnosed (e.g <5 years) Type 2 diabetics Qatar residents with a body mass index (BMI) of >30.0 to <40.0 kg/m2
  Interventions: Behavioral: 10-week exercise programme based on aerobic interval and resistance training

INTERVENTIONS:
Behavioral: 10-week exercise programme based on aerobic interval and resistance training — The intervention will take place over 10 weeks. Participants will complete three sessions per week; each sessions will be scheduled at least 24 hours apart. Two sessions per week will consist of aerobic interval exercise and resistance training, and one session per week will consist of aerobic interval exercise only.

SUMMARY:
The prevalence of type 2 diabetes (T2DM) is increasing sharply around the world and obesity and sedentary lifestyles are driving the epidemic. Obesity is often, but not always present in patients with T2DM. The primary aim of this study is to understand the impact of the ratio of lean body mass (metabolically active skeletal muscle) to adipose tissue mass on the severity of insulin resistance and pancreatic beta cell dysfunction in non-obese and obese Qatar residents with T2DM. An exercise programme aimed to increase lean mass and aerobic capacity will be initiated for a period 10 weeks in non-obese and obese early onset diabetics who are residents of Qatar. The effect of the exercise programme on total body fat, regional fat distribution and intramuscular and intrahepatic fat content using magnetic resonance imaging (MRI) in these groups of diabetics will be assessed and related to total body insulin sensitivity and β-cell function as measured with the gold standard methods: the euglycemic clamp technique and arginine stimulation. Genetic approaches including candidate gene testing and non-targeted miRNA expression profiling and metabolomics are employed. Physical fitness pre- and post-intervention will also be assessed. The impact of the exercise programme on conventional inflammatory markers, the phenotype of immune cells, metabolic hormones, and markers of oxidative stress, endoplasmic reticulum stress and heat shock response (Hsp-72, Hsp -40/DNAJB3 and Hsp-25) are studied in relation to metabolic changes. Through this study, the contributions of fitness, fatness and exercise training on insulin resistance and beta cell function will be elucidated in Qatari residents with T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. New onset T2DM (<5 years duration).
2. Aged 18 and 60 years.
3. Residents of Qatar with intention to stay for the duration of the study (approx 4 months)
4. Otherwise healthy or with stable, treated medical conditions (hypertension, hyperlipidemia, hypothyroidism, etc.)
5. Hemoglobin A1c (HbA1c) level < 8%.
6. "Diet and lifestyle" or metformin or DPP4 inhibitors prescribed for T2DM.
7. Willingness and ability to comply with the exercise protocol and study duration.

Exclusion Criteria:

1. Type 1 Diabetes Mellitus or history of hospitalization for hyperglycemia or suspected ketoacidosis.
2. T2DM prescribed insulin, or any other anti-diabetic agent other than metformin or DDP4 inhibitors.
3. HbA1c ≥8.0%.
4. Body mass index (BMI) ≤ 18.5 kg/m2 (underweight) and ≥ 40 kg/m2 (morbid obese).
5. Reported weight loss or gain (± 2 kg) over the preceding three months;
6. Pregnant or lactating women or women planning to be pregnant during the course of the study.
7. History of regular exercise (the equivalent of 150 minutes of moderate intensity aerobic and/or 2 sessions of resistance training per week) or of a job that demands a similar degree of physical activity within the past 6 months.
8. Use of medications that affect glucose metabolism, glucose tolerance or body weight including oral corticosteroids and atypical anti-psychotics.
9. History of cardiovascular disease including previous myocardial infarction, congestive cardiac failure, valvular heart disease, stroke or the use of medication to alter coagulation including daily aspirin, anti-platelet drugs or any class of anticoagulant or a clinically significant abnormality on electrocardiogram that in the opinion of a consulting cardiologist should prevent participation.
10. History of chronic diseases associated with inflammation and/or the daily use of anti-inflammatory or immunosuppressant medications for arthritis, gout, rheumatologic disorders, inflammatory bowel disease, or viral infections including hepatitis B, C and HIV.
11. History of psychiatric disorders including current clinical depression, schizophrenia, bipolar disorder or subjects with known claustrophobia.
12. History of chronic neurological disorders such as epilepsy, dementia or movement disorders.
13. Hematocrit <33%.
14. Participation in other research studies that require blood drawing or any medical, nutritional or behavioral intervention.
15. The presence of large ferromagnetic tattoos that may interfere with the MRI determination of body fat.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 10 weeks
  Insulin sensitivity will be assessed using a modification of the De Fronzo technique 2-hour Euglycemic Clamp procedure.

SECONDARY OUTCOMES:
Glucose regulation/ insulin sensitivity | 10 weeks
  Glucose regulation and insulin sensitivity will be assessed via a 4-hour Oral glucose tolerance test procedure.
Pancreatic beta-cell function | 10 weeks
  Pancreatic beta-cell function will be assessed using a 3-hour Arginine stimulation test procedure.
Hepatic insulin resistance index | 10 weeks
  The measurement of hepatic insulin resistance index will completed during euglycemic clamp procedure.
Vascular reactivity | 10 weeks
  Endothelial reactivity will be assessed during the euglycemic clamp procedure, using an standard blood pressure arm cuff and the VENDYS instrument.
Body Mass Index (BMI) | 10 weeks
  Patient's weight and height will be measured in kilograms (kg) and meters (m), respectively, and combined to report BMI in kg/m^2
Body fat profiling | 10 weeks
  Mesenteric, hepatic, subcutaneous and skeletal muscle infiltrating fat will be measured with a 3.0T MR-scanner using a whole-body Dixon protocol. Hepatic fat content and skeletal muscle fat infiltration will be measured. All measurements will be performed with 3T Phillips Ingenia scanner.
Total body fat | 10 weeks
  Dual energy X-ray absorptiometry (DEXA), via the Lunar iDXA instrument and enCORE software will be used to derive total body fat.
Non-fat mass | 10 weeks
  Dual energy X-ray absorptiometry (DEXA), via the Lunar iDXA instrument and enCORE software will be used to derive non-fat mass.
Visceral adipose volume | 10 weeks
  Dual energy X-ray absorptiometry (DEXA), via the Lunar iDXA instrument and enCORE software will be used to derive estimates of visceral adipose volume.
Cardiorespiratory fitness (estimated maximal oxygen uptake) | 10 weeks
  Maximal oxygen uptake (VO2max) will be estimated using the Astrand and Rhyming cycle ergometer protocol.
Upper body strength | 10 weeks
  Upper body strength will be determined via handgrip strength using a handgrip dynanmometer. Assessments will be conducted on both hands.
Physical function | 10 weeks
  Physical function will be measured using the 6-minute walk test.
Lower body strength | 10 weeks
  Lower body strength will be assessed using the 30-s sit to stand test.
Fasting Plasma glucose | 10 weeks
  The number of particiapnts that have improvement in fasting plasma glucose.

OTHER OUTCOMES:
Heart rate during exercise sessions | 10 weeks
  Heart rate will be recorded using polar H10 monitors and the polar team system throughout exercise programme.

CONTACTS AND LOCATIONS:
Overall Officials: Monica C Skarulis, MD, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar